CLINICAL TRIAL: NCT00001342
Title: A Study of Collateral Disorders of Glycogen Storage Disease
Brief Title: Study of Glycogen Storage Disease and Associated Disorders
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 930020; 93-CH-0020
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-10

CONDITIONS: Glycogen Storage Disease
Keywords: Electrooculography; Electroretinogram; Fluorescein Angiogram; Glycogen Storage Disease
MeSH Terms: conditions — Glycogen Storage Disease

SUMMARY:
Glycogen, is the storage form of glucose. It is usually formed from sugar and stored in the liver. When tissues, such as muscle, need glucose for fuel the stored glycogen is converted into glucose with the help of enzymes produced in the body. Glycogen storage disease (GSD) refers to a group of conditions characterized by abnormal storage of glycogen due to the absence of particular enzymes needed in the process of storing and using glycogen.

This study addresses the related metabolic abnormalities of glycogen storage disease (GSD). As patients with disorders of glycogen metabolism are followed it becomes apparent that the condition is much more complex than initially thought.

Researchers believe that patients suffering from glycogen storage disorders should be followed and monitored for other heritable metabolic disorders.

This study will attempt to determine the frequency of associated disorders in patients with GSD. In addition, the study will look at the current management of these patients to see if the prognosis and course of the disease is changed.

DETAILED DESCRIPTION:
This study addresses the related metabolic abnormalities of the glycogeneses. As more older individuals with glycogen storage disease are followed and studied, it becomes apparent that when individuals with glycogenosis are viewed from a longitudinal perspective, the condition is much more complex and diverse in its related conditions than one would have reason to believe, even in hindsight. It is relevant to follow these individuals, searching for abnormalities not only with glycogen storage disease in mind, but also because other heritable metabolic disorders, including cystinosis and cystic fibrosis, reflect the accumulation of associated disorders with age which often have no apparent direct association with GSD.

ELIGIBILITY:
Patients age 20 or older, male or female.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20
Dates: Start 1992-11; Study Completion 2001-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), Bethesda, Maryland, United States

REFERENCES:
- [Background] Chen YT, Coleman RA, Scheinman JI, Kolbeck PC, Sidbury JB. Renal disease in type I glycogen storage disease. N Engl J Med. 1988 Jan 7;318(1):7-11. doi: 10.1056/NEJM198801073180102. PMID 3422104
- [Background] Goans RE, Weiss GH, Vieira NE, Sidbury JB, Abrams SA, Yergey AL. Calcium kinetics in glycogen storage disease type 1a. Calcif Tissue Int. 1996 Dec;59(6):449-53. doi: 10.1007/BF00369209. PMID 8939770